CLINICAL TRIAL: NCT06597097
Title: Evaluation of Interprofessional Relations Between Primary Care and Hospital Centers in the Experimentation of Medical Cannabis in France Carried Out by the ANSM
Brief Title: Evaluation of Interprofessional Relations Between Primary Care and Hospital Centers in the Experimentation of Medical Cannabis in France Carried Out by the ANSM (ECIPCanna)
Acronym: ECIPCanna
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0215
Record Dates: First submitted 2024-04-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Medical Cannabis
Keywords: Cannabis for medical use; Outpatient medicine; Prescription; Pharmacy; Primary care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study to explore inter-professional relations and perceptions around the experimentation of medical cannabis, conducted by the French National Agency for Safety and Health. The study aims to identify the barriers and facilitators to prescribing and dispensing medical cannabis and to analyse healthcare professionals' perceptions of medical cannabis in France. Using a qualitative method based on semi-directed interviews and focus groups, the study will involve hospital physicians, general practitioners, and community and hospital pharmacists participating in the the French National Agency for Safety and Health experiment. The primary objective is to understand the dynamics between health professionals involved in the medical cannabis programme, while secondary objectives include proposing strategies to overcome barriers to the provision of medical cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professional participating in the experiment conducted by the the French National Agency for Safety and Health: Hospital doctor, general practitioner, community pharmacist, or hospital pharmacist
* Non-opposition

Exclusion Criteria:

* Refusal of participation by hospital doctor, general practitioner, community pharmacist, or hospital pharmacist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals participating in the experiment conducted by the French National Agency for Safety and Health:
  * Hospital doctors
  * General practitioners
  * Community pharmacists
  * Hospital pharmacists
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Exploring the inter-professional relationships of those involved in the medical cannabis experiment being conducted by the French National Agency for Safety and Health | 1 day
  Construct mental maps of representations relating to the prescription and dispensing of medical cannabis.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement